CLINICAL TRIAL: NCT03652233
Title: Afatinib and Nivolumab for Treatment of Recurrent/Metastatic Squamous Cell Carcinoma of the Head and Neck (SCCHN) Not Previously Treated With Immunotherapy.
Brief Title: Afatinib and Nivolumab as Treatment for Recurrent/Metastatic Squamous Cell Carcinoma of the Head and Neck
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Comprehensive Cancer Network (Network); Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Michael K. Gibson, Principal Investigator, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC HN 1840; NCI-2018-01790 (Registry Identifier: NCI, Clinical Trials Reporting Program)
Record Dates: First submitted 2018-08-20; First posted 2018-08-29 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Recurrent Squamous Cell Carcinoma of the Head or Neck; Metastatic Squamous Cell Carcinoma of the Head or Neck; Squamous Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Squamous Cell | interventions — Nivolumab; Afatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Afatinib and Nivolumab (Experimental)
  Interventions: Drug: Nivolumab; Drug: Afatinib

INTERVENTIONS:
Drug: Nivolumab — Given by vein every 14 days for up to 12 months
Drug: Afatinib — Taken by mouth daily for up to 12 months

SUMMARY:
This phase I/Ib trial will assess the dose, safety and side effects of the combination of the cancer drugs afatinib (GILOTRIF®) and nivolumab (OPDIVO®) and to assess the anti-cancer effects of this combination of drugs when used to treat patients with advanced head and neck cancers that did not respond to previous treatments.

DETAILED DESCRIPTION:
Primary Objectives:

Phase I: To determine dose limiting toxicities (DLTs) and maximum tolerated dose (MTD) of afatinib when given in combination with nivolumab for subjects with recurrent/metastatic Squamous Cell Carcinoma of the Head and Neck not previously treated with immunotherapy

Phase IB: To determine long term safety of afatinib in combination with nivolumab when administered to subjects with recurrent/metastatic Squamous Cell Carcinoma of the Head and Neck who had experienced disease progression during or after platinum- and cetuximab-based chemotherapy regimen.

Secondary Objectives:

To assess progression free survival and overall survival of afatinib in combination with nivolumab when given to subjects with recurrent/metastatic Squamous Cell Carcinoma of the Head and Neck not previously treated with immunotherapy.

To estimate HPV stratified ORR as assessed by irRECIST in recurrent/metastatic Squamous Cell Carcinoma of the Head and Neck not previously treated with immunotherapy.

Exploratory Objectives:

* Determination of key molecular alterations that may confer treatment resistance. Specifically, we will examine key somatic mutations in ERBB1 (exons 18-21), ERBB2 (exon 20), and BRAF (V600) genes. We will further characterize the expression levels of ErbB2 and phosphatase and tensin homolog (PTEN) in tumor samples.
* Characterization of active CD8+ T-cell density and PD-L1 expression levels in the tumor parenchyma pre- and on-treatment. Immunogenicity will be assessed by expression and localization of key molecules PD-1, PD-L1, CTLA-4, TIM-3, LAG-3 and OX40 within the tumor parenchyma.
* Characterization of circulating monocytic myeloid-derived suppressor cells (m-MDSCs) frequency from pre-treatment peripheral blood samples.
* Characterization of HBD3 expression in the tumor parenchyma from pre-treatment tumor tissue samples.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent/metastatic Squamous Cell Carcinoma of the Head and Neck not previously treated with immunotherapy
* No prior immunotherapy for this disease, including therapies targeting PD-

  1, PD-L1, CTLA-4 or other cells and molecules aiming to modulate immune response against Squamous Cell Carcinoma of the Head and Neck.
* ECOG Performance Status of 0-1
* Normal organ and marrow function as defined below:

  * WBC ≥ 2000 cells/μL
  * Absolute neutrophil count (ANC) ≥ 1000 cells/μL
  * Hemoglobin (Hgb) ≥ 9 g/dL
  * Platelets ≥ 100,000/μL
  * Estimated creatinine clearance ≥ 30 ml/min
  * Left ventricular function with resting ejection fraction ≥ 50%
  * Total bilirubin < 1.5 X ULN (Subjects with Gilbert's syndrome total bilirubin must be ≤4 times institutional upper limit of normal)
  * AST and ALT of < 2.5 X ULN
* Ability to understand and the willingness to sign a written informed consent document.
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to the start of Nivolumab. WOCBP must use appropriate method(s) of contraception. WOCBP should use an adequate method to avoid pregnancy for 23 weeks (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug.
* Recovered from any previous therapy related toxicity to ≤ Grade 1 at study entry (except for stable sensory neuropathy ≤ Grade 2 and alopecia).
* Availability of a "newly obtained" standard of care biopsy obtained through either core or excisional biopsy. A newly obtained sample may be obtained up to 28 days prior to treatment initiation. Tissue beyond the 28-day window may be considered with the approval Protocol Chair. Tissue that has been previously irradiated or surgically intervened is acceptable

Exclusion Criteria:

* Currently receiving any other investigational agents or using an investigational agent 30 days prior to the first dose of trial treatment.
* Disease that is suitable for local therapy with curative intent.
* Untreated brain metastases/CNS disease excluded because of poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Subjects with stable, treated CNS metastases are eligible.
* Known hypersensitivity to afatinib or nivolumab.
* Prior EGFR-targeted small molecule therapy except cetuximab.
* Hormonal therapy with the exception of those used for diabetes or birth control is not allowed.
* Radiotherapy within 4 weeks prior to randomization, except as follows:

Palliative radiation to target organs other than chest may be allowed up to 2 weeks prior to randomisation, and Single dose palliative treatment for symptomatic metastasis outside above allowance to be discussed with sponsor prior to enrolling.

* Major surgery within 4 weeks before starting study treatment or scheduled for surgery during the projected course of the study.
* History or presence of clinically relevant cardiovascular abnormalities such as uncontrolled hypertension (systolic blood pressure ≥ 160 or diastolic blood pressure ≥ 90), congestive heart failure NYHA classification of ≥ 3, unstable angina or poorly controlled arrhythmia as determined by the investigator. Myocardial infarction within 6 months prior to the enrollment.
* Previous or concomitant malignancies at other sites, except effectively treated non-melanoma skin cancers, carcinoma in situ of the cervix, ductal carcinoma in situ or effectively treated malignancy that has been in remission for more than 3 years and is considered to be cured.
* Requiring treatment with any of the prohibited concomitant medications listed in section 6.4 that cannot be stopped for the duration of trial participation.
* Known active or pre-existing interstitial lung disease.
* Any history or presence of poorly controlled gastrointestinal disorders that could affect the absorption of the study drug (e.g. Crohn's disease, ulcerative colitis, chronic diarrhea and malabsorption).
* Prior immune checkpoint targeted therapy, including anti-PD-1, anti-PD-L1 or anti-PD-L2.
* History of autoimmune disease or disease requiring immunosuppression therapy.
* Uncontrolled inter-current illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Women must not be breastfeeding.
* Men who are sexually active with WOCBP must use any contraceptive method (Appendix II) with a failure rate of less than 1% per year Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 31 weeks after the last dose of investigational product Women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile as well as azoospermic men do not require contraception.
* Testing positive Human Immunodeficiency Virus (HIV) acquired immunodeficiency syndrome (AIDS).
* Active hepatitis B or hepatitis C.
* Active infection requiring systemic antibiotic treatment or intensive care.
* Active non-infectious pneumonitis
* Received live vaccine within 30 days of start of study treatment.
* Known psychiatric or substance abuse disorders that may interfere with cooperation with the requirements of the trial.
* Other significant medical conditions that may interfere with surgical biopsy and afatinib and nivolumab administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-11-02 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (phase I) | Up to 42 days
Dose limiting toxicities (phase I) | Up to 42 days
Number of participants with treatment-related adverse events as assessed by CTCAE version 4.0 | Up to 24 months

SECONDARY OUTCOMES:
Progression free survival | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years
Overall survival | From date of enrollment to date of death from any cause assessed up to 3 years.
Objective response rate | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Mike Gibson, MD, PhD, Principal Investigator — Vanderbilt-Ingram Cancer Center